CLINICAL TRIAL: NCT00179179
Title: The Effects of Nutrition Supplementation and Resistance Exercise During Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50189; R01DK045604 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dietary Supplements; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): nutritional supplement plus resistance exercise
  Interventions: Drug: nutritional supplementation; Behavioral: exercise
- 2 (Active Comparator): nutritional supplement only (resistance exercise will not be performed)
  Interventions: Drug: nutritional supplementation

INTERVENTIONS:
Drug: nutritional supplementation — 2 oral ingestions per study visit of protein supplement containing a total of 960 kilocalories: 132.8 kilocalories from protein, 412.8 kilocalories from carbohydrates, and 412.8 kilocalories from fat; 6 study visits over a 12-month period
Behavioral: exercise — resistance training on a duel leg press consisting of 3 sets of 8-12 repetitions; the first 5 study visits over a 12-month period
  Arms: 1

SUMMARY:
To test the hypothesis that an exercise session combined with adequate nutritional supplementation improves skeletal muscle protein accretion during a hemodialysis session.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis for more than 3 months, on a thrice weekly hemodialysis program.
* Adequately dialyzed (Kt/V > 1.2).
* Age 18-75

Exclusion Criteria:

* Pregnant women.
* Patients unable to perform exercise
* Severe unstable underlying disease besides commonly associated with ESRD. Cardiac patients that are stable will be included.
* Patients hospitalized within the last month prior to the study.
* Patients with malfunctioning arterial-venous access (recirculation and/or blood flow < 750 ml/min)
* Patients receiving steroids and/or other immunosuppressive agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
improvement in net protein muscle balance | 10 hours

SECONDARY OUTCOMES:
improvement in net whole body protein balance | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States